CLINICAL TRIAL: NCT04865848
Title: Comparison of Articaine Mandibular Infiltration to Lidocaine Inferior Alveolar Nerve Block in Pediatric Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: research operation issues
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Evelina Hristova Kratunova, Clinical Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-0160
Record Dates: First submitted 2020-05-14; First posted 2021-04-29 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia
Keywords: Lidocaine; Articaine; Children; Dental; Local; Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandibular infiltration dental anesthesia with Articaine (Experimental): Step-by-step:
  * Reflect tissue to expose injection site.
  * Orient bevel of the needle to be parallel to the bone and insert needle into mucobuccal fold
  * Proceed to the depth that approximates the apices of the buccal roots of the primary molars.
  * Aspirate.
  * Deposit bolus of local anesthetic slowly at a rate of 1 ml/min.
  * Remove needle.
  * A subsequent lingual infiltration is delivered.
  The armamentarium includes: 4% articaine HCl with 1:100,000 epinephrine (Septocaine ®, Septodont, Lancaster, Penn. USA) in 1.7 ml cartridges and 30-gauge short needle manufactured by Henry Schein® (Melville, N.Y., USA). All injections are given using a self-aspirating syringe (A-Titan, Orchard Park, N.Y., USA).
  Interventions: Procedure: Dental local anesthesia
- Inferior Alveolar Nerve Block with Lidocaine (Active Comparator): Step-by-step:
  * Dry injection site with gauze.
  * The barrel of the syringe should be directed on a plane between the two primary molars on the opposite side of the arch. It is advisable to inject a small amount of the solution as soon as the tissue is penetrated and to continue to inject minute quantities as the needle is directed toward the mandibular foramen.
  Insert to the depth that is adjacent to bone.
  * Aspirate.
  * Slowly inject bolus of anesthetic at a rate of 1 ml/min.
  * Remove needle.
  The armamentarium includes 2% lidocaine HCl with 1:100,000 epinephrine (Henry Schein ® Lidocaine, Novocol, Cambridge, Ontario, Canada) in 1.7 ml cartridges, as well as 27-gauge long needles manufactured by Henry Schein® (Melville, N.Y., USA). All injections are given using a self-aspirating syringe (A-Titan, Orchard Park, N.Y., USA).
  Interventions: Procedure: Dental local anesthesia

INTERVENTIONS:
Procedure: Dental local anesthesia — Dental local anesthesia

SUMMARY:
This is a prospective, single-blind, parallel-design randomized controlled clinical trial that aims compare the effectiveness of articaine local infiltration to lidocaine inferior alveolar nerve block (IANB) for restorative treatment of primary mandibular molars (PMM). Four to 10-year-old children who needed PMM restorations are enrolled according to inclusion criteria and randomly allocated into the articaine or lidocaine group. One operator administers all local anesthesia (LA). Using the Modified Behavioral Pain Scale, 15 trained and calibrated examiners, blinded to LA type, evaluate the subjects' reactions during LA administration and treatment. Children rate their experience using the Wong-Baker FACES Pain Rating Scale. Subjects' blood pressure and pulse throughout the visit are recorded. Results are statistically analyzed using independent t-tests, Mann Whitney-U, and Repeated Measures ANOVA (P<0.05).

DETAILED DESCRIPTION:
This is a parallel design randomized controlled trial that aims to evaluate the effectiveness of mandibular infiltration anesthesia with Articaine in comparison to IANB with Lidocaine used for restorative and pulp therapy procedures in pediatric patients.

Lidocaine (2% Lidocaine Hydrochloride with 1:100,000 Epinephrine) and Articaine (4% Articaine Hydrochloride with 1:100,000 Epinephrine) are compared and evaluated for their effectiveness of anesthetizing primary mandibular molars for restorative and pulp therapy procedures. A number of clinical and behavioral variables including blood pressure, pulse, physical movements, and pain perception are evaluated.

Participants for this study will be recruited from the pool of patients attending the Post-graduate (PG) clinic at the Pediatric Dentistry Department of the College of Dentistry (COD), University of Illinois at Chicago (UIC). Inclusion and exclusion criteria are specified separately for the selected patients and for the teeth involved. Informed consent from the parent/guardian and assent from the pediatric participant (7 years of age and older) will be obtained and signed. This is a prospective randomized clinical trial utilizing a random digit table for participant allocation into either the Articaine Group or the Lidocaine Group. The dosage of LA will be determined by the child's body weight and will not exceed the maximum recommended 4.4 mg/kg for Lidocaine and 7 mg/kg for Articaine. Before the injection, 20% Benzocaine topical anesthetic gel will be applied at the injection site with a cotton swab for approximately 3 minutes over dry mucosa. The randomly assigned LA, either Lidocaine IANB or Articaine infiltration, will be administered. One designated operator, an experienced specialist pediatric dentist, will conduct all LA injections to all participants. A trained and calibrated dental assistant (examiner A) will record the child's reactions during the LA administration using the Modified Behavioral Pain Scale (MBPS), adapted by Taddio et al. 1994. This scale allows for objective evaluation of pain using multiple criteria such as facial display, movement of extremities, movement of torso, and crying. A second trained and calibrated investigator (examiner B), a resident in pediatric dentistry, who is blinded to the type of LA agent used, will complete the planned dental treatment for the primary mandibular molars. Examiner B will complete MBPS (#B) evaluating the patient's reactions during the dental treatment. Generally, effective LA results in less negative and more positive patient's reactions to the dental care. In total, 15 examiners A and 17 examiners B will take part in the study. All examiners will be trained and calibrated with respect to the use of MBPS. During the entire treatment visit, each participant will wear a pulse and blood pressure monitor. The machine will produce automatic recordings every 10 minutes. Patients that experience distress and pain can exhibit increased pulse and blood pressure values outside of the considered normal range per age. At the end of the dental visit, the pediatric patient will be asked to complete a Wong-Baker FACES® Pain Response Scale (PRS) for feedback of their experience with the entire dental visit. The PRS contains six images of varying facial expression ranging from laughter to tears which are assigned at numerical value for objective evaluation. All used data will be coded and captured on specifically designed for the purposes of the study evaluation forms. The data gathered through all study forms will be transferred into Microsoft® Excel 2018 and the statistical analysis will be carried out with IBM SPSS Statistics.

ELIGIBILITY:
Inclusion Criteria:

Per patient:

* Medical status: ASA I: a normal, healthy patient;
* Age range: from 4 to 10 year old patients (males and females);
* Past history of dental treatment using local anesthetic;
* Cooperative for dental treatment (Frankel 3 or 4);
* Obtained informed consent to participate in the study;
* English speakers;

B. Per tooth:

• Primary mandibular molar; Tooth that requires restorative dental care, including intracoronal or extracoronal restorations, due to:

* Caries;
* Pulp treatment (indirect pulp therapy, pulpotomy, or pulpectomy);
* Developmental defects;
* Tooth surface loss (erosion/attrition);

Exclusion Criteria:

A. Per patient:

* Medical status: patients in category II,III, IV, V, VI of the ASA physical status classification system:
* Age: younger than 4 years of age or older than 10 years of age;
* No history of dental treatment using local anesthetic;
* Uncooperative for dental treatment (Frankel 1 or 2);
* Informed consent to participate in the study not obtained;
* Non-English speakers;

B. Per tooth:

* Tooth other than mandibular primary molar
* Tooth requiring extraction

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Effectiveness of articaine local infiltration to lidocaine inferior alveolar nerve block (IANB) for restorative treatment of primary mandibular molars (PMM). | up to 24 hour later (as the parent is able to contact the principal investigator and report any issues). Numerical value of 0 is assigned to the cases that did not report any adverse events and a numerical value of 1 to reported adverse outcomes.
  The primary outcome measure for this study is to compare the effectiveness of articaine local infiltration to lidocaine inferior alveolar nerve block (IANB) for restorative treatment of primary mandibular molars (PMM).

SECONDARY OUTCOMES:
Secondary outcome measures | Immediately after procedure
  Pain assessment will be conducted using the Modified Behavioral Pain Scale (MBPS), which measures infant pain during immunizations based on facial expression, cry, and bodily movements. Scores range from 0 to 10, comparable to the visual analog scale (VAS) for child pain assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Evelina Kratunova, Principal Investigator — University of Illinois at Chicago
Locations (1):
- College of Dentistry, Univesity of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No